CLINICAL TRIAL: NCT01521312
Title: A Randomized, Double Blind, Placebo Controlled, Pilot Study to Evaluate ACute and Chronic Effects of Saxagliptin on Impaired Glucose Tolerance and micro-and Macro-vascular Integrators
Brief Title: ACute and Chronic Effects of Saxagliptin
Acronym: ACCES
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P101105
Record Dates: First submitted 2011-11-22; First posted 2012-01-30 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-01

CONDITIONS: Impaired Glucose Tolerance
Keywords: Impaired glucose tolerance; Saxagliptin; Cardiovascular risk integrators; Vago-sympathetic activity; Arterial stiffness; Endothelial function
MeSH Terms: conditions — Glucose Intolerance | interventions — saxagliptin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saxagliptin (Experimental): Saxagliptin 5 mg (tablet) at BREAKFEAST
  Interventions: Drug: saxagliptin
- placebo pill (Placebo Comparator): at BREAKFEAST
  Interventions: Other: placebo pill

INTERVENTIONS:
Drug: saxagliptin — 5mg a day for 11-14 weeks
  Other Names: Onglyza
  Arms: Saxagliptin
Other: placebo pill — one tablet a day for 11-14 weeks
  Arms: placebo pill

SUMMARY:
Glucose ACCES study will explore the acute and long term (12-week treatment) effects of saxagliptin in patients with impaired glucose tolerance during fasting and after a standardised breakfast. The investigations will be performed on:

* glycemic parameters
* on cardiovascular parameters

DETAILED DESCRIPTION:
The aim of this pilot study is to compare in patients with impaired glucose tolerance the effects of saxagliptin versus placebo:

(i) on glucose metabolism (ii) on vago-sympathetic activity, arterial stiffness and endothelial function. A total of 36 patients will be recruited in the department of Endocrinology-Diabetology-Nutrition of Jean VERDIER hospital, AP-HP, Bondy, France.

The measurements will be performed in the morning 1) at the time of randomisation (Acute ACCES study) and 2) 11-14 weeks after the beginning of saxagliptin or placebo (Chronic ACCES study).

We will evaluate at fasting and each hour after a standardized breakfast:

(i) biological and metabolic parameters. Furthermore, an oral glucose tolerance test will be performed at the end of the study.

(ii) by non-invasive devices arterial stiffness (Sphygmocor®), endothelial function (ENDOPAT 2000® ), cutaneous microcirculation (laser doppler Perimed ®.PF 5010) and cardiac autonomic function(task force monitor®).

ELIGIBILITY:
Inclusion Criteria:

* Social security affiliation
* Persons without TUTORSHIP that can freely agree to participate to the study
* Age between 18 to 70 years
* Impaired glucose tolerance diagnosed during the previous month.

Exclusion criteria:

* Pregnancy
* Breast feeding
* Diabetes
* No contraception
* Body Mass Index > 45 kg/m²
* Arterial blood pressure > 160/110 mmHg
* Creatinine clearance < 60 ml/min
* Severe hepatocellular insufficiency
* Chronic respiratory disease
* Anaemia (Hemoglobin < 10 g/dl)
* Peripheral arterial occlusive disease
* Heart failure
* Cardiac arrhythmia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Vago-sympathetic activity. | First day (inclusion) and after 11-14 weeks of treatment
  This is a pilot study. The vascular measurements will be performed before and during a standardized breakfast.
arterial stiffness | First day (inclusion) and after 11-14 weeks of treatment
  This is a pilot study. The vascular measurements will be performed before and during a standardized breakfast.
endothelial function | First day (inclusion) and after 11-14 weeks of treatment
  This is a pilot study. The vascular measurements will be performed before and during a standardized breakfast.
oral glucose tolerance test. | First day (inclusion) and after 11-14 weeks of treatment
  This is a pilot study. The vascular measurements will be performed before and during a standardized breakfast.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Valensi, MD, Principal Investigator — Jean Verdier Hospital - Department of Endocrinology-Diabetology-Nutrition
Locations (1):
- Jean Verdier hospital, Department of Endocrinology-Diabetology-Nutrition, Bondy, France

REFERENCES:
- [Derived] Rezki A, Cosson E, Fysekidis M, Chiheb S, Vicaut E, Valensi P. Acute and long-term effects of saxagliptin on a set of cardiovascular targets measured at fasting and post-prandially in obese patients with impaired glucose tolerance: A placebo-controlled study. Nutr Metab Cardiovasc Dis. 2021 Sep 22;31(10):2945-2958. doi: 10.1016/j.numecd.2021.06.017. Epub 2021 Jul 1. PMID 34420816
- [Derived] Rezki A, Fysekidis M, Chiheb S, Vicaut E, Cosson E, Valensi P. Acute and long-term effects of saxagliptin on post-prandial glycemic response in obese patients with impaired glucose tolerance. Nutr Metab Cardiovasc Dis. 2021 Apr 9;31(4):1257-1266. doi: 10.1016/j.numecd.2020.12.025. Epub 2020 Dec 31. PMID 33618922